CLINICAL TRIAL: NCT04191785
Title: Evaluation of the Plasmatic and Urinary Neutrophil Gelatinase - Associated Lipocalin as a Predictive Marker of Renal Injury in Children With Febrile Urinary Infection
Brief Title: Evaluation of the Plasmatic NGAL as a Predictive Marker of Renal Injury in Children With Urinary Infection. (Perf-NGAL-IU)
Acronym: Perf-NGAL-IU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-HPNCL-08
Record Dates: First submitted 2019-08-27; First posted 2019-12-10 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- plasmatic NGAL and MRI (Experimental)
  Interventions: Diagnostic Test: plasmatic NGAl and MRI

INTERVENTIONS:
Diagnostic Test: plasmatic NGAl and MRI — Determination of plasma NGAL protein during routine blood test Realization of a reno vesical MRI at 48 hours of inclusion

SUMMARY:
Urinary infections in children is very common. Delay in the diagnosis may be followed by complications.

Pyelonephritis is a febrile urinary infection with a renal injury. In local experience, about 30-40% of the children don't have an inflammatory syndrome or echographical abnormalities. Do they really have a renal injury ? In fact, only the scintigraphy or the Magnetic Resonance Imaging (MRI) may show these lesions, but are done only in specific cases (diagnosis of uropathy or nephropathy). Recent studies have shown that plasmatic Neutrophil Gelatinase-Associated Lipocalin (NGAL) is associated traumatic or inflammatory renal lesions. But the plasmatic NGAL cutoff is fluctuant depending on the cohorts and gold standards. The main goal is to evaluate a new methodology of dosing NGAL, (immuno-dosage turbidimetric dosage). The investigators suppose that plasmatic NGAL protein will detect renal injury, which would be confirmed by MRI.

The aim of this study is to evaluate the area under the curve (AUC) of plasmatic NGAL protein with an automatised method, for the detection of renal injury. This would be confirmed by reno vesical MRI, in children over 2 years old with febrile urinary infections

DETAILED DESCRIPTION:
Urinary infections in children is very common and should be diagnosed as soon as possible. Delay in the diagnosis ma be followed by complications such as sepsis, renal scar, high blood pressure, renal insufficiency.

The diagnosis may be tough when it comes to children because of its unspecific symptomatology. Pyelonephritis is a febrile urinary infection associated to renal abnormalities. Following the french recommendations ("Sociéte de Pathologie Infectieuse de Langue Française" The French Society of Infectious disease SPILF and "Groupe de Pathologies Infectieuses Pédiatriques" The Pediatric infectious disease Group GPIP 2015), the investigators should first use an intravenous probabilistic antibiotic during minimum 48 hours to lower the bacterial inoculum. Then, the investigators should switch to an oral antibiotic during 8 days to sterilise the urines.

In local experience, about 30 to 40 % of the children don't have an inflammatory syndrom or echographical abnormalities. Do they really have a renal injury? In fact, only the scintigraphy or the Magnetic Resonance Imaging (MRI) may show these lesions, but are done only in specific cases (diagnosis of uropathy or nephropathy). Recent studies have shown that plasmatic Neutrophil Gelatinase-Associated Lipocalin (NGAL) is associated traumatic or inflammatory renal lesions. But the plasmatic NGAL cutoff is fluctuant depending on the cohorts and gold standards. In those studies, dosing NGAL was non automatised and long.

the investigators would like to evaluate a new methodology of dosing NGAL, (immuno-dosage turbidimetric dosage). The investigators suppose that plasmatic NGAL protein will detect renal injury, which would be confirmed by MRI.

This is an interventional, prospective, multicentered study. It will last for 2 years. The aim of this study is to evaluate the AUC of plasmatic NGAL protein with an automatised method, for the detection of renal injury. This would be confirmed by reno vesical MRI, in children over 2 years old with febrile urinary infections.

ELIGIBILITY:
Inclusion Criteria:

* Children over 4 years old, continent
* Fever ≥ 38,5 degrés Celsius for less than 4 days
* Positive urine strip
* Parental authorisation
* Using french Health Care System

Exclusion Criteria:

* Uropathy
* 2nd febrile urinary infection
* No parental authorisation
* Non confirmed Urinary infection on a well done Cyto Bacteriological Urine (CBU)
* Urinal contamination defined by : ≥ 2 bacterial, urinal bacteriuria < 10^5 Colony Forming Unit (CFU)/ml

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Compare plasmatic Neutrophil Gelatinase-Associated Lipocalin (NGAL) with gold standard Reno vesical Magnetic Resonance Imaging (MRI) | 48 hours after inclusion
  NGAL will be evaluated in urines, and plasma. The method will be automatised. The dosage will be from 25 to 5000 ng/ml. Gold standard will be MRI (nephritis is defined by hyperintense zones in diffusion sequence and hyposignal in ADC mode)
  The primary outcome measure is to estimate the area under the curve (AUC) defining the different measures of the performance (Sensitivity, specificity) of plasmatic NGAL protein in ng/ml according to the presence or not of a kidney lesion diagnosed at the RMI (gold standard).

SECONDARY OUTCOMES:
Define performance of plasmatic NGAL for the diagnostic of renal abnormality due to a pyelonephritis | 48 hours after inclusion
  The performance of NGAL will be evaluated (sensitivity, specificity, positive predictive value, negative predictive value) using the chosen cutoff of NGAL. Gold standard will be reno vesical MRI
Performance and area under the curve (AUC) of C-reactive Protein (CRP) for the diagnostic of pyelonephritis | 48 hours after inclusion
  The performance (sensitivity, specificity, positive predictive value, negative predictive value) and the AUC of CRP will be defined using the following cutoff (CRP > 20 mg/l ) chosen from the litterature. CRP will be dosed by an automatised method on XL Siemens machine.
Performance and area under the curve (AUC) of Procalcitonin (PCT) for the diagnostic of pyelonephritis | 48 hours after inclusion
  The performance (sensitivity, specificity, positive predictive value, negative predictive value) and the AUC of PCT will be defined using the following cutoff ( PCT > 0,5 ng/ml) chosen from the litterature. PCT will be dosed using a Brahms automat
Compare the AUC of plasmatic NGAL and CRP | 48 hours after inclusion
  AUC for plasmatic NGAL will be compared to AUC of CRP, AUC will be calculated using receiver operator characteristic (ROC) curves
Compare the AUC of plasmatic NGAL and PCT. | 48 hours after inclusion
  AUC for plasmatic NGAL will be compared to AUC of PCT. AUC will be calculated using receiver operator characteristic (ROC) curves
Performance of urinary NGAL | 48 hours after inclusion
  Define an area under receiver operator characteristic (ROC) curve based on the dosage of urinary NGAL used to diagnose renal abnormality. The method will be automatised. The dosage will be from 25 to 5000 ng/ml. Gold standard will be MRI (nephritis is defined by hyperintense zones in diffusion sequence and hyposignal in Apparent Diffusion coefficient (ADC) mode).
Performance of doppler echography | 48 hours after inclusion
  The performance of doppler echography (sensitivity, specificity, positive predictive value, negative predictive value) will be established using MRI as a gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Tran Antoine, MD, Principal Investigator — Children Hopital of Nice CHU-Lenval Emergency
Locations (1):
- Fondation Lenval Hopitaux Pediatriques de Nice Chu Lenval, Nice, France